CLINICAL TRIAL: NCT04953598
Title: Ultrasonic Measurement of the Area of the Anterior Superior Labrum of the Hip Joint for Diagnosis of Labrum Tear
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018106
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Acetabular Labrum Tear
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acetabular labrum tears: Patients with clinically diagnosed acetabular labrum tears
  Interventions: Diagnostic Test: Ultrasonography
- Patients with non-hip injuries: For non-hip joint reasons, come to the ultrasound department of our hospital to diagnose patients at the same time, and exclude other past and current hip diseases
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Patient undergoes diagnostic ultrasound examination

SUMMARY:
In this study, ultrasound diagnosis was performed for patients with hip joint anterior superior labrum tear, and the final surgical observation was used as the gold standard to evaluate the diagnostic efficacy of ultrasonic measurement of the hip joint anterior superior labrum area in the diagnosis of labrum tear.

DETAILED DESCRIPTION:
In this study, ultrasound diagnosis was performed for patients with a torn anterior superior labrum of the hip joint, and the final surgical observation was the gold standard. The control group selected patients with non-hip joint reasons to come to the ultrasound department of our hospital for diagnosis at the same time. Both the case group and the control group were included in the study at a rate of 1.1 times. This study plans to include 149 cases in the case group and 297 cases in the control group. This study was used to evaluate the diagnostic efficacy of ultrasonic measurement of the area of the anterior superior labrum of the hip in the diagnosis of labrum tears.

ELIGIBILITY:
Inclusion Criteria:

Case group inclusion criteria (1) Age is greater than or equal to 18 years old (2) Patients with preoperative ultrasound examination for clinically planned hip joint anterior superior labrum tear (3) The patient can understand and sign the informed consent form Control group inclusion criteria

1. Age is greater than or equal to 18 years old
2. Patients who come to the ultrasound department of our hospital for treatment of non-hip joints at the same time
3. The patient can understand and sign the informed consent form

Exclusion Criteria:

Case group exclusion criteria

1. Mental conditions are not allowed
2. Adhesives that are allergic to any known Control group exclusion criteria

(1) Mental conditions are not allowed (2) Adhesives that are allergic to any known (3) Past and current diseases of other hip joint diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case group: Outpatient Department of Sports Medicine, Peking University Third Hospital, clinically diagnosed patients with hip joint labrum tear, preoperative ultrasound examination.
  Control group: Patients who came to our hospital's ultrasound department at the same time for non-hip joint reasons matched by age, gender and case group.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-07-29 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Ultrasound diagnosis result image | ultrasound diagnosis were preformed with hip arthroscopy at the same 1 day visiting time point
  Ultrasound diagnosis as hip joint anterior superior labrum tear

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Cui, Study Chair — Peking University Third Hospital
Locations (1):
- Department of Ultrasound Diagnosis, Peking University Third Hospital, Beijing, Beijing Municipality, China